CLINICAL TRIAL: NCT06729190
Title: Combined Effect of Biofeedback and Functional Electrical Stimulation on Upper Limb Functions in Children With Hemiplegia
Brief Title: Effect of Biofeedback and Functional Electrical Stimulation in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Eldin Taha Ramadan, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/005003
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator): Physical therapy program The exercise session for one hour for each child , conducted 3times/ week for 3 successive months.
  1. Flexibility exercises for shorted muscles and spastic muscles.
  2. Strengthening training focusing on the trunk lower limb and upper limb muscles for weak muscles.
  3. Postural control exercise in different positions and different surfaces
  4. General endurance training
  5. Exercises to facilitate hand function
  6. Exercises included, grasping a cube, transferring cube, removing and placing pegs, releasing cube and placing cubes. Strengthening exercises of the intrinsic muscles of the hand
  Interventions: Procedure: Physical therapy program
- Group B (Experimental): The exercise session for one hour for each child same as group A, conducted 3times/ week for 3 successive months plus the combined biofeedback therapy and FES at anti spastic muscles (shoulders flexors, elbow and wrist extensors
  Interventions: Device: biofeedback; Procedure: Physical therapy program

INTERVENTIONS:
Device: biofeedback — biofeedback therapy and FES at anti spastic muscles(shoulders flexors, elbow and wrist extensors) while doing specific exercises (including basic reaching, grasping, carrying, release
  Arms: Group B
Procedure: Physical therapy program — Flexibility exercises for shorted muscles and spastic muscles, Strengthening training focusing on the trunk lower limb and upper limb muscles for weak muscles, Postural control exercise in different positions and different surfaces, General endurance training, Exercises to facilitate hand function, Exercises included, grasping a cube, transferring cube, removing and placing pegs, releasing cube and placing cubes. Strengthening exercises of the intrinsic muscles of the hand

SUMMARY:
40 children with hemiplegia cerebral palsy from both sex will be recruited from outpatient clinic of abo resh hospital ,their age ranged from 5-10 years

DETAILED DESCRIPTION:
40 children with hemiplegia cerebral palsy from both sex will be recruited ,their age ranged from 5-10 years, treatment includes functional electrical nerve stimulation and biofeedback to assess their combined effect on upper limb function

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 5 to 10 years.
* Spasticity grade range from 1+ to 2, according to Modified Ashworth Scale (MAS) (Bohannon and Smith, 2011).
* Their UL ability function will be at level II according to Manual Ability Classification System (MACS) (Penta et al., 2001).
* They will be able to follow instructions.

Exclusion Criteria:

* Loss of sensation
* The presence of visual or auditory impairments.
* Musculoskeletal problems or fixed deformities in the upper extremities.
* Seizures.
* Surgical interference in upper limbs.
* Botulinum toxin injections in the last 6 months.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
hand function in children with CP | pre intervention and re assessed after 3 months of treatment
  hand function in children with CP will be assessed by The Quality of Upper Extremity Skills Test

SECONDARY OUTCOMES:
Range of motion | pre intervention and re assessed after 3 months of treatment
  Range of motion will be assessed using Electronic goniometer
muscle grip strength | pre intervention and re assessed after 3 months of treatment
  muscle grip strength will be assessed using Hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A Mamdouh, PHD, Study Director — professor of physical therapy; Eman I Alhadedy, PHD, Study Director — Professor of physical therapy; Amira I Fathi, Study Director — Lecturer of physical therapy
Locations (1):
- Cairo University, Giza, Egypt